CLINICAL TRIAL: NCT01436084
Title: Phase II Study of SB1518 for Patients With Myelodysplastic Syndrome (MDS)
Brief Title: SB1518 for Patients With Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Colloborating sponsor decision.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0427
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndrome; MDS; SB1518
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB1518 (Experimental): 400 mg orally a day for 28 day cycle.
  Interventions: Drug: SB1518

INTERVENTIONS:
Drug: SB1518 — 400 mg taken orally, once daily without regard of food, 28 day cycle.

SUMMARY:
The goal of this clinical research study is to learn if SB1518 can help to control myelodysplastic syndrome. The safety of the drug will also be studied.

SB1518 is designed to block JAK2 and FLT3. SB1518 may have anti-tumor activity in certain leukemias, myelofibrosis, and lymphoma.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take SB1518 by mouth 1 time every day. You can take it with or without food, and it should be taken at the same time every day.

You will receive your monthly supply of SB1518 during your clinic visit. The capsules should not be opened or crushed. Do not touch the powder in the capsules. If you do, wash effected areas thoroughly with water.

Each study cycle is 28 days.

Study Visits:

At every study visit, you will be asked about any drugs you may be taking, and any side effects you have had.

One (1) time a week during Cycle 1, blood (about 2 tablespoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond, blood (about 2 tablespoons) will be collected for routine tests.

On Day 28 of each cycle, you will have a bone marrow aspirate and/or biopsy to check the status of the disease. If the screening bone marrow test showed unusual genetic test results, these samples will be used for cytogenetic testing. If you have a response to therapy, you will have a bone marrow aspirate and/or biopsy every 3 cycles, if your doctor thinks it needed.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, you are able to undergo allogeneic bone marrow transplantation, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit.

End-of-Treatment Visit:

At 30 days after your last dose of study drug, you will have an end-of-treatment visit.

* You will be asked about any drugs you may be taking, and any side effects you have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspirate and/or biopsy to check the status of the disease, if your doctor thinks it is needed.

This is an investigational study. SB1518 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 40 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS by the IPSS classification including low, int-1, int-2, and high risk are eligible. Patients should have received at least one line of prior therapy including growth factors, lenalidomide, or hypomethylating agents.
2. Signed informed consent.
3. Age >/= 18 years old.
4. Patients must have the following non-hematologic values: Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) </= 2.5 x Upper Limit of Normal (ULN) if both are available or </= 5.0 x ULN if hepatic involvement is present as determined by the investigator; Serum bilirubin </=2 x ULN; Serum creatinine </= 2 x ULN or 24-hour creatinine clearance >/= 50 ml/min
5. Patients, if sexually active, must agree to use appropriate forms birth control.

Exclusion Criteria:

1. Uncontrolled intercurrent illness, including but not limited to ongoing active infection or psychiatric illness or social situations that the treating physician judges would limit compliance with study requirements. Patients receiving antibiotics for infections that are under control may be included in the study.
2. History of myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure within 6 months prior to study enrollment;
3. New York Heart Association Class III or IV congestive heart failure;
4. Ongoing cardiac dysrhythmias of Grade >/= 2, atrial fibrillation of any grade, QTc prolongation > 470 ms or other factors that increase the risk of QT prolongation (e.g., heart failure; hypokalemia, defined as serum potassium < 3.0 mEq/L; family history of long QT interval syndrome);
5. Required use of a concomitant medication known to prolong the QT interval significantly.
6. Known HIV seropositivity;
7. Known active hepatitis A, B, or C;
8. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 22, 2011 to January 24, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Four participants of the eight enrolled failed to meet the screening criteria and were not treated on the study. The study was closed to new patient entry 2 months after activation due to sponsor/collaborator issues; the only patient remaining was taken off study at that time.
Period: Overall Study
Arm/Group | SB1518
Started | 4
Completed | 0
Not Completed | 4
Not completed — Disease Progression | 2
Not completed — Withdrawal by Subject | 1
Not completed — Early Closure of Study | 1

BASELINE CHARACTERISTICS:
Arm/Group | SB1518
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 69 [57 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Overall response based on hematologic improvement defined by International Working Group (IWG) response criteria in myelodysplasia. Complete remission (CR): Bone marrow of 5% myeloblasts with normal maturation of all cell lines, noted persistent dysplasia; Partial Remission: CR criteria if abnormal before treatment except Bone marrow blasts decreased by 50% over pretreatment but still > 5%; Marrow CR: Bone marrow 5% myeloblasts and decrease by 50% over pretreatment. Bone marrow aspirate pre-therapy (Day 0) and on Day 28 of first cycle then every 3 cycles. Responses must last at least 4 weeks.
Time Frame: 28 days to one year
Population: Study was halted prior to completion of treatment and assessment for any participant(s).
Arm/Group | SB1518
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected during 28 day drug cycles to thirty days following the last dose of study drug. In the absence of treatment delays due to adverse events, treatment may continue indefinitely. Study period December 2011 to January 2012.
Arm/Group | SB1518
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB1518 (N=4)
Abdominal pain (General disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Gastrointestinal (GI) Other (Gastrointestinal disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Pain Other (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No